CLINICAL TRIAL: NCT00738920
Title: Self Administered CBT for IBS: A Multisite Trial
Brief Title: Self Administered Cognitive Behavior Therapy for Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Northwestern University Feinberg School of Medicine (Other); Frontier Science & Technology Research Foundation, Inc. (Industry); RTI International (Other)
Responsible Party: Principal Investigator, Jeffrey Lackner, Principal investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DK77738; U01DK077738 (NIH)
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Results first posted 2022-07-06 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-07

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MC-CBT (Active Comparator): Self Administered Cognitive Behavior Therapy
  Interventions: Behavioral: Self Administered Cognitive Behavior Therapy
- Standard-CBT (Active Comparator): Therapist Administered Cognitive Behavior Therapy
  Interventions: Behavioral: Therapist Administered Cognitive Behavior Therapy
- Education/Support (Active Comparator): Behavioral Patient Education/Counseling
  Interventions: Behavioral: Behavioral Education and Supportive Therapy

INTERVENTIONS:
Behavioral: Self Administered Cognitive Behavior Therapy — This 4 session treatment is aimed at controlling symptoms by changing specific behaviors found to aggravate IBS
  Arms: MC-CBT
Behavioral: Therapist Administered Cognitive Behavior Therapy — This 10 session treatment is aimed at controlling symptoms by changing specific behaviors found to aggravate IBS
  Arms: Standard-CBT
Behavioral: Behavioral Education and Supportive Therapy — This 4 session treatment aims at controlling symptoms through support and the provision of information about IBS symptoms, how it is diagnosed, its causes, and treatment options and a collaborative, relationship between the patient and doctor
  Arms: Education/Support

SUMMARY:
The primary goal of the proposed trial is to assess the short- and long-term efficacy of cognitive behavior therapy (CBT) for irritable bowel syndrome using two treatment delivery systems (self administered, therapist administered). Secondary aims seek to specify the conditions under which CBT may (or may not) achieve its effects (moderator questions), why and how these effects are achieved (mediator questions) and at what economic cost. Long term project goals are to develop an effective self-administered behavioral treatment program that can enhance the quality of patient care, improve clinical outcomes, and decrease the economic and personal costs of one of the most prevalent and intractable GI disorders.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a chronic, prevalent, often disabling, GI disorder for which there is no reliable and satisfactory medical option for its full range of symptoms (abdominal pain, bowel dysfunction). An accumulating body of evidence indicates that a specific psychosocial treatment called cognitive behavioral therapy (CBT) is associated with significant reductions in IBS symptoms and related difficulties. Despite its apparent efficacy, CBT's clinical effectiveness (i.e., its generalizability, feasibility, cost effectiveness) has not been adequately established due partly to its duration, cost, and limited accessibility. As the "second generation" of IBS treatments undergo development and validation, it has become increasingly clear that efficacy demonstration is a necessary but not sufficient condition of treatment viability. In a pilot study funded under NIDDK's R03 mechanism, we addressed these problems by developing a briefer, largely self administered version of CBT that requires only 4, 1 hr clinic visits. Our RCT data showed that a 10 session version of CBT can be translated into a 4 session version without compromising patient acceptability or short term efficacy. It is unclear whether treatment effects are maintained long term (out to 12 months), due to theoretical change mechanisms (vs. nonspecific factors common across different forms of therapy), are more pronounced among specific subgroups of patients, or, generalize to a large sample of Rome III diagnosed patients treated by different investigative sites. We seek to address these questions by conducting a larger, more definitive, multisite RCT that will recruit from 2 treatment sites 480 patients with moderate to severe IBS and assess their acute and long term response to brief (4 session) CBT, extended (10 session) CBT, or a credible education/support condition. We will use the first year to develop a clinical infrastructure to ensure the success and integrity of the proposed trial. In the short term, a successful trial will lend empirical validation to a self administered version of CBT that retains the efficacy of standard CBT but is more transportable, accessible to patients outside of research protocols, and less costly to deliver. In the long term, we hope to show that a self guided behavioral treatment program is an effective and efficient treatment delivery system that can enhance the quality of patient care, improve clinical outcomes, and decrease the economic and personal costs of one of the most prevalent and intractable GI disorders.

ELIGIBILITY:
Inclusion Criteria:

* Males or female patients aged 18 to 70 years (inclusive);
* All ethnic groups;
* Meet Rome III criteria for IBS with symptoms of at least moderate severity (at least 2 days per week);
* Ability to understand and provide informed consent;
* With the exception of antibiotics, participant is willing to remain on a stable dose only through the 4-week pretreatment baseline period prior to randomization;
* Participant either not taking medications or if taking medications willing to suspend starting any new medications only during the initial 4-week pretreatment baseline period;
* Participant demonstrates an ability to speak understand and read, English a the sixth grade level or higher;
* Willingness to be randomized to CBT or Support/Education to which s/he has been assigned to to adhere to protocol requirements;
* Participant is willing to attend regularly scheduled therapy session during active phase of the trial;
* Participant is willing to be contacted and scheduled for follow-up assessment at week 12 and 3, 6, 9, and 12 months after the conclusion of acute treatment phase;
* Participant is willing and able to enter symptom information into an assigned portable computer and complete questionnaires through treatment and at regularly scheduled follow ups
* Participant has access to a telephone; and
* Participant is willing and able to provide adequate information for locator purposes.

Exclusion Criteria:

* Evidence of current structural or biochemical abnormalities or medication use that better explain the participant's IBS symptoms (e.g. IBD);
* Evidence of a current infection or infection of any type within the 2 weeks prior to the study gastroenterologists' evaluation which would obscure the presentation of IBS symptoms. In such cases the baseline can be delayed until 2 weeks after complete recovery.
* Participant has received antibiotics (e.g. rifaximin and or neomycin) specifically targeted to treat IBS symptoms within the past 3 months. In this instance eligibility will be suspended for 12 weeks from the initial date the antibiotic was consumed.
* Participant has undergone previous abdominal surgery that would have caused significant alternation of the anatomy/physiology of the digestive/GI tract, which adequately explains GI symptoms;
* Participant has been diagnosed and/or treated for malignancy in the past 5 years with the exception of localized basal or squamous cell carcinomas of the skin;
* Participant has an unstable extraintestinal medical condition whose immediate or foreseeable treatment needs (e.g., hospitalization, conflicting physician visits) would realistically interfere with study demands (e.g., consistent attendance at treatment sessions and/or ability to participate in telephone interventions) or may affect the interpretation of clinical efficacy data;
* Participant has a major psychiatric disorder, which in the opinion of the senior clinical staff may impede conduct of the clinical trial. These disorders include but are not limited to major depression diagnosis with a high risk of suicidal behavior (i.e. intent or plan), alcohol or substance abuse/dependence within the past year, a lifetime history of schizophrenia or schizoaffective disorder or gross cognitive impairments;
* Participant has other conditions which in the opinion of the senior clinical staff would influence negatively the conduct of the clinical trial;
* Participant is currently receiving targeted psychotherapy for IBS and is unwilling or unable to discontinue his/her treatment for the acute treatment phase of this study;
* Participant is unable to complete all scheduled screening visits; and participant is inaccessible for interventions and/or follow-up evaluations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2010-08; Primary Completion 2016-12 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lackner, PsyD, Principal Investigator — State University of New York at Buffalo; Laurie Keefer, Ph.D., Principal Investigator — Ichan School of Medicine at Mount Sinai; Jeffrey Lackner, Psy.D., Study Chair — State University of New York at Buffalo
Locations (2):
- United States (2):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University at Buffalo School of Medicine, Buffalo, New York

IPD SHARING:
Plan to Share IPD: Yes
One of the main goals of the IBSOS is to establish a central repository of data for subsequent hypothesis-based research designed to enable the widest dissemination of data, while also protecting the privacy of the participants and the utility of the data by de-identification and masking of potentially sensitive data elements. To support these objectives we will catalog and provide basic results sets through the NIDDK repository www.niddkrepository.org, as well as create and deliver more comprehensive de-identified data sets, for each completed aim of the IBSOS study. Study data will be provided in SAS/SPSS format and will be named to match corresponding codebooks or dictionary and study forms, which will also be located within the Repository. Codebooks will include variable names and labels, where applicable. For analysis data sets, we will provide documentation for analyses conducted for manuscript publication as well as descriptive summaries for main variables.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Baseline data: September 1, 2018 Primary outcome manuscript: May 1, 2018 Entire dataset from intervention study: September 1, 2019
Access Criteria: All applications for access of these data sets must be submitted through an application to NIDDK central repository as outlined on their website www.niddkrepository.org. Access for the data submitted to the NIDDK Data Repository will be determined by the NIDDK. All investigators who receive IBSOS resources must agree to acknowledge the IBSOS Study and the NIDDK central repository.

REFERENCES:
- [Derived] Jacobs JP, Gupta A, Bhatt RR, Brawer J, Gao K, Tillisch K, Lagishetty V, Firth R, Gudleski GD, Ellingson BM, Labus JS, Naliboff BD, Lackner JM, Mayer EA. Cognitive behavioral therapy for irritable bowel syndrome induces bidirectional alterations in the brain-gut-microbiome axis associated with gastrointestinal symptom improvement. Microbiome. 2021 Nov 30;9(1):236. doi: 10.1186/s40168-021-01188-6. PMID 34847963
- [Derived] Lackner JM, Jaccard J, Keefer L, Brenner DM, Firth RS, Gudleski GD, Hamilton FA, Katz LA, Krasner SS, Ma CX, Radziwon CD, Sitrin MD. Improvement in Gastrointestinal Symptoms After Cognitive Behavior Therapy for Refractory Irritable Bowel Syndrome. Gastroenterology. 2018 Jul;155(1):47-57. doi: 10.1053/j.gastro.2018.03.063. Epub 2018 Apr 25. PMID 29702118
- [Derived] Lackner JM, Keefer L, Jaccard J, Firth R, Brenner D, Bratten J, Dunlap LJ, Ma C, Byroads M; IBSOS Research Group. The Irritable Bowel Syndrome Outcome Study (IBSOS): rationale and design of a randomized, placebo-controlled trial with 12 month follow up of self- versus clinician-administered CBT for moderate to severe irritable bowel syndrome. Contemp Clin Trials. 2012 Nov;33(6):1293-310. doi: 10.1016/j.cct.2012.07.013. Epub 2012 Jul 28. PMID 22846389

RESULTS

PARTICIPANT FLOW:
Period: Baseline to 2-Week Follow-Up
Arm/Group | MC-CBT | Standard-CBT | Education/Support
Started | 145 | 146 | 145
Completed | 129 | 123 | 130
Not Completed | 16 | 23 | 15
Not completed — Lost to Follow-up | 8 | 9 | 8
Not completed — Withdrawal by Subject | 8 | 14 | 7
Period: 2-Week Follow-Up to 3-Month Follow-Up
Arm/Group | MC-CBT | Standard-CBT | Education/Support
Started | 129 | 123 | 130
Completed | 121 | 111 | 118
Not Completed | 8 | 12 | 12
Not completed — Withdrawal by Subject | 3 | 5 | 6
Not completed — Lost to Follow-up | 5 | 7 | 6
Period: 3-Month Follow-Up to 6-Month Follow-Up
Arm/Group | MC-CBT | Standard-CBT | Education/Support
Started | 121 | 111 | 118
Completed | 117 | 111 | 115
Not Completed | 4 | 0 | 3
Not completed — Lost to Follow-up | 3 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1
Period: 6-Month Follow-Up to 9-Month Follow-Up
Arm/Group | MC-CBT | Standard-CBT | Education/Support
Started | 117 | 111 | 115
Completed | 113 | 104 | 103
Not Completed | 4 | 7 | 12
Not completed — Lost to Follow-up | 2 | 4 | 7
Not completed — Withdrawal by Subject | 2 | 3 | 5
Period: 9-Month Follow-Up to 12-Month Follow-Up
Arm/Group | MC-CBT | Standard-CBT | Education/Support
Started | 113 | 104 | 103
Completed | 112 | 103 | 102
Not Completed | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MC-CBT | Standard-CBT | Education/Support | Total
Number analyzed (Participants) | 145 | 146 | 145 | 436
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (14.6) | 41.1 (14.4) | 42.2 (15.4) | 41.4 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 112 | 114 | 350
  Male | 21 | 34 | 31 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 7 | 7 | 9 | 23
  White | 131 | 127 | 125 | 383
  More than one race | 4 | 4 | 6 | 14
  Unknown or Not Reported | 1 | 4 | 3 | 8
Predominant IBS Bowel Type [Count of Participants; unit: Participants]
  Constipation | 43 | 40 | 47 | 130
  Diarrhea | 59 | 67 | 62 | 188
  Mixed | 33 | 35 | 30 | 98
  Undifferentiated | 10 | 4 | 6 | 20
Duration of IBS symptoms [Mean (Standard Deviation); unit: years] | 15.7 (13.3) | 17.7 (13.3) | 17.7 (16.4) | 17.1 (14.4)
Medication Use for IBS Symptoms [Count of Participants; unit: Participants]
  Pain medication | 9 | 13 | 13 | 35
  Bowel medication | 86 | 87 | 98 | 271
  Multisymptom medication | 6 | 7 | 7 | 20
  Psychiatric medication | 8 | 12 | 6 | 26
  None | 36 | 27 | 21 | 84

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impressions - Improvement Scale (CGI-I; Patient Version)
Description: The CGI-I is a single-item, 7-point centered scale that integrates symptom severity and improvement since the start of treatment. Specific IBS-based anchor points were used, as is the convention for multi-symptom disease states. Response range from 1 (very much worse) to 7 (very much improved), with higher scores indicating greater symptom improvement. Participants who respond 6 (much improved) or 7 (very much improved) are classified as treatment responders.
Time Frame: 2-Week Follow-Up, 3-Month Follow-Up, 6-Month Follow-Up, 9-Month Follow-Up and 12-Month Follow-Up
Population: Per protocol
Measure: Number; unit: percentage of treatment responders
Arm/Group | MC-CBT | Standard-CBT | Education/Support
Number analyzed (Participants) | 131 | 125 | 133
percentage of treatment responders
  2-Week Follow-Up: number analyzed (Participants) | 129 | 123 | 130
  2-Week Follow-Up | 68.1 | 64.6 | 46.7
  3-Month Follow-Up: number analyzed (Participants) | 121 | 111 | 118
  3-Month Follow-Up | 64.0 | 64.6 | 49.5
  6-Month Follow-Up: number analyzed (Participants) | 117 | 111 | 115
  6-Month Follow-Up | 63.9 | 58.1 | 51.0
  9-Month Follow-Up: number analyzed (Participants) | 113 | 104 | 103
  9-Month Follow-Up | 64.9 | 62.2 | 48.9
  12-Month Follow-Up: number analyzed (Participants) | 112 | 103 | 102
  12-Month Follow-Up | 70.0 | 68.4 | 51.7

2. Secondary Outcome: Change From Baseline on the IBS Symptom Severity Scale (IBS-SSS)
Description: The IBS-SSS is a 5-item instrument used to measure severity of abdominal pain, frequency of abdominal pain, severity of abdominal distention, dissatisfaction with bowel habits, and interference with QOL. For four of the items, respondents mark a point on a 101 mm visual analogue scale to indicate their response to that item. The proportional distance from zero is the score (ranging from 0 to 100) assigned for that scale. The other item asks the number of days out of 10 the patient experiences abdominal pain and the answer is multiplied by 10 to create a 0 to 100 metric. The five items are summed and the total scores range from 0-500, with higher scores signifying more severe symptoms [mild (<175), moderate (175-300), severe (>300)]. A decrease of 50 points on the IBS-SSS is considered clinically significant.
Time Frame: Baseline, 2-Week Follow-Up, 3-Month Follow-Up, 6-Month Follow-Up, 9-Month Follow-Up and 12-Month Follow-Up
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MC-CBT | Standard-CBT | Education/Support
Number analyzed (Participants) | 131 | 125 | 133
units on a scale
  Change from Baseline to 2-Week Follow-Up: number analyzed (Participants) | 129 | 123 | 130
  Change from Baseline to 2-Week Follow-Up | -89.4 (17.0) | 81.0 (17.0) | 84.4 (14.6)
  Change from Baseline to 3-Month Follow-Up: number analyzed (Participants) | 121 | 111 | 118
  Change from Baseline to 3-Month Follow-Up | -105.9 (17.7) | -103.2 (16.4) | -88.5 (14.6)
  Change from Baseline to 6-Month Follow-Up: number analyzed (Participants) | 117 | 111 | 115
  Change from Baseline to 6-Month Follow-Up | -111.3 (17.9) | -103.5 (17.7) | -97.93 (15.4)
  Change from Baseline to 9-Month Follow-Up: number analyzed (Participants) | 113 | 104 | 103
  Change from Baseline to 9-Month Follow-Up | -111.2 (17.7) | -104.6 (17.0) | -94.9 (17.1)
  Change from Baseline to 12-Month Follow-Up: number analyzed (Participants) | 112 | 103 | 102
  Change from Baseline to 12-Month Follow-Up | -120.1 (17.9) | -112.9 (18.4) | -103.4 (18.6)

3. Secondary Outcome: Client Satisfaction Questionnaire (CSQ)
Description: The CSQ is an 8-item questionnaire that measures patient satisfaction with treatment. Scores range from 8 to 32 with higher scores indicating greater satisfaction with treatment.
Time Frame: 2-Week Follow-Up
Population: Per protocol
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MC-CBT | Standard-CBT | Education/Support
Number analyzed (Participants) | 129 | 123 | 130
units on a scale | 28.9 [28.3 to 29.5] | 28.4 [27.7 to 29.1] | 26.6 [25.7 to 27.5]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | MC-CBT | Standard-CBT | Education/Support
All-Cause Mortality (participants affected / at risk) | 0/145 | 0/146 | 0/145
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/146 | 1/145
Other Adverse Events (participants affected / at risk) | 0/145 | 0/146 | 0/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MC-CBT (N=145) | Standard-CBT (N=146) | Education/Support (N=145)
Attempted suicide (Social circumstances) | 0 | 0 | 1 (1) — Attempted suicide with no reasonable possible relationship to intervention. Resolved with sequelae.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No